CLINICAL TRIAL: NCT00622570
Title: Comparison of Effectiveness of Pentobarbital and Thiopental in Patients With Refractory Intracranial Hypertension.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slowly recruitment rate. Intermediate analysis
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Dr. Jon Pérez Bárcena, Hospital Son Dureta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 02/0642; IB
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2007-07

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury, barbiturate coma
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Pentobarbital; Thiopental

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pentobarbital
  Interventions: Drug: Pentobarbital
- 2 (Active Comparator): thiopental
  Interventions: Drug: thiopental

INTERVENTIONS:
Drug: Pentobarbital — 10 mg/kg in 30 minutes; then 5 mg/kg/h during 3 hours; then 1 mg/kg/h
  Other Names: Nembutal(r)
  Arms: 1
Drug: thiopental — 2 mg/kg in bolus; if ICP is not below 20 mmHg then 3 mg/kg in bolus; if ICP is not below 20 mmHg it can be administrated a third bolus of 5 mg/kg.
  Maintenance: 3 mg/kg/h in perfusion
  Other Names: PENTOTHAL(R)
  Arms: 2

SUMMARY:
Objective: to assess the effectiveness of pentobarbital and thiopental to control raised intracranial pressure (ICP), refractory to first level measures, in patients with severe traumatic brain injury.

Material and methods: prospective, randomized open study to compare the effectiveness between two treatments: pentobarbital and thiopental. The patients will be selected from those admitted to the Intensive Care Unit with a severe traumatic brain injury (postresuscitation Glasgow Coma Scale equal or less than 8 points) and raised ICP (ICP>20 mmHg) refractory to first level measures according to the Brain Trauma Foundation guidelines. The adverse effects of both treatments were also collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a severe closed head injury and a post-resuscitation Glasgow Coma Scale (GCS) score below or equal to 8
* Age between 15 and 76 years (inclusive)
* High ICP (> 20 mm Hg) refractory to first-tier therapeutic measures according to BTF guidelines (1)
* Hemodynamic stability defined as a systolic blood pressure of at least 100 mm Hg or above at the moment of entering the trial
* Written informed consent obtained from next-of-kin or the patient's legally authorized representative

Exclusion Criteria:

* Previously known ischemic heart failure (Ejection fraction < 35%)
* Pregnancy
* bilateral dilated and unreactive pupils and a GCS of 3
* Intolerance to barbiturates

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-05; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Intracranial pressure control | along intensive care unit stay

SECONDARY OUTCOMES:
Hypotension (Mean arterial blood pressure<80 mmHg) | during barbiturate treatment
Infection | during barbiturate treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jon Perez, MD, Principal Investigator — Son Dureta Hospital
Locations (1):
- Son Dureta Hospital, Palma, Balearic Island, Spain

REFERENCES:
- [Result] Perez-Barcena J, Barcelo B, Homar J, Abadal JM, Molina FJ, de la Pena A, Sahuquillo J, Ibanez J. [Comparison of the effectiveness of pentobarbital and thiopental in patients with refractory intracranial hypertension. Preliminary report of 20 patients]. Neurocirugia (Astur). 2005 Feb;16(1):5-12; discussion 12-3. Spanish. PMID 15756405
- [Derived] Perez-Barcena J, Llompart-Pou JA, Homar J, Abadal JM, Raurich JM, Frontera G, Brell M, Ibanez J, Ibanez J. Pentobarbital versus thiopental in the treatment of refractory intracranial hypertension in patients with traumatic brain injury: a randomized controlled trial. Crit Care. 2008;12(4):R112. doi: 10.1186/cc6999. Epub 2008 Aug 29. PMID 18759980